CLINICAL TRIAL: NCT00205439
Title: Fluorescence Bronchoscopic Surveillance For New Lung Primaries After Curative Therapy for Squamous Cell Carcinoma of the Aerodigestive Tract"
Brief Title: Surveillance For New Lung Primaries
Status: Terminated | Type: Observational
Why Stopped: low accrual
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: CC01506; 2001-431 (Other: Institutional Review Board)
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2019-11-15 (Actual); Status verified 2015-07

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

GROUPS / COHORTS (1):
- Fluorescence bronchosopy with sputum cytology: Patients undergo surgery with Fluorescence bronchosopy and sputum cytology.

SUMMARY:
The primary goal of this study is to determine the prevalence of tracheobronchial carcinomas in patients with a history of squamous cell cancer of the aerodigestive tract who have been treated with a curative intent and remain disease free. Detection of pre-invasive and invasive lesions (moderate to severe dysplasia, CIS) with fluorescence bronchoscopic surveillance may help to define the natural history of these lesions and allow earlier intervention should they progress to invasive lesions.

ELIGIBILITY:
Inclusion Criteria:

* History squamous cell NSCLC who have undergone complete resection or definitive chemotherapy

Exclusion Criteria:

* History of an aerodigestive tract carcinoma of non-squamous histology
* Patients who have Stage IIIA, IIIB or IV squamous cell lung cancer that have undergone resection or chemotherapy within three years
* Patients who have Stage I or II squamous cell lung cancer that have undergone resection or chemotherapy within one year
* Patients who have received external beam radiation therapy for treatment of a squamous cell cancer of the lung

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with new lung primaries after curative therapy for squamous cell carcinoma of the aerodigestive tract
Enrollment: 200 (Estimated)
Dates: Start 2001-12; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tracey Weigel, MD, Principal Investigator — University of Wisconsin Medical School
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/